CLINICAL TRIAL: NCT05572424
Title: Interest of an Adapted Physical Activity (APA) Program Among Patients With Juvenile Idiopathic Arthritis: a Feasibility and Efficacy Preliminary Study
Acronym: ATHLETIQUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/600
Record Dates: First submitted 2022-07-25; First posted 2022-10-07 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Glutamyl Aminopeptidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptated Physical Activity + pedometer watch (Experimental): Follow an Adapted Physical Activity program during 12 weeks and wear a pedometer watch during 1 year
  Interventions: Other: Adaptated Physical Activity (APA) + pedometer watch
- Control group (No Intervention): Usual care

INTERVENTIONS:
Other: Adaptated Physical Activity (APA) + pedometer watch — Adapted physical activities program : 12 weeks, 2 40-minutes sessions per week ( one broadcast live via online video conferencing and other one in autonomy according to a sequence of different personalized exercises defined by the APA's professional). Children are divided into 6 groups. Each session will be broken down into three parts: the warm-up (10mins), the session's corps alternating between five to eight of muscle strengthening, proprioception, and endurance exercises (20mins) and a cool-down with stretching (10mins). The physical activity performed during the sessions will be quantified with a heart rate monitor and the range of 60-70% of the maximum theoretical heart rate for each child will be respected.
  A pedometer watch will wear during 1 year and will provide the number of steps.
  Arms: Adaptated Physical Activity + pedometer watch

SUMMARY:
The Juvenile Idiopathic Arthritis (JIA) affects joints mobility and leads pain, impacting the practice of physical activities. Adapted Physical Activities are rehabilitation methods increasingly used, but additional studies are needed to define the nature of the physical activity for patients with JIA. The ATHLETIQUE project aims to evaluate the impact of a program integrating APA sessions together with the wearing of a pedometer watch on disease activity of patients with JIA.

ELIGIBILITY:
Inclusion criteria:

* Children (boys and girls) aged 6 to 17 years
* Children with juvenile idiopathic arthritis (JIA) : oligoarticular, polyarticular, psoriatic or enthesitis-related arthritis, with more than one year of disease progression
* Children on stable conventional or biotherapy 3 months prior to inclusion
* Children with a computer/tablet/connected phone that allows them to follow adapted physical activities sessions online
* If sexually active adolescents, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double barrier method, contraceptive patches)
* Signed informed consent to participate indicating that the parent(s) understand the purpose and procedures required for the study and agree(s) that their child(ren) will participate in the study and abide by the requirements and restrictions of the study
* Affiliation with a French social security system or beneficiary of such a system.

Non-inclusion criteria:

* Treatment by intra-articular infiltration less than 1 month old (immobilization required after the procedure and temporary cessation of physical activity unavoidable)
* Contraindications to physical activity
* Subject unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant adolescent
* Subject in the exclusion period of another study or is the "national volunteer register"

Exclusion criteria :

* Intra-articular infiltration treatment during the 3 months of the adapted physical activity (APA) program (except for the temporomandibular joint)
* Change of biotherapy during the 3 months of the APA program if the treatment is ineffective
* Physical inability to engage in physical activity, unrelated to JIA, during the 3-month of the APA program

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Juvenile Arthritis Disease Activity-27 Score Assesment | Week 14
  JADAS-27 score includes 4 components :
  1. number of inflammatory joints among 27 joints identified,
  2. a medical assesment of clinical disease activity with Visual Analogic Scale (from 0 point = worst to 10 points = best),
  3. assesment of assesment of patient's well-being by the patient or a parent with Visual Analogic Scale (froom 0 point = worst to 10 points = best),
  4. sedimentation rate (from 0 to 10).

SECONDARY OUTCOMES:
Juvenile Arthritis Disease Activity-27 Score Assesment | Weeks 26 and 50
  JADAS-27 score includes 4 components :
  1. number of inflammatory joints among 27 joints identified,
  2. a medical assesment of clinical disease activity with Visual Analogic Scale (from 0 point = worst to 10 points = best),
  3. assesment of assesment of patient's well-being by the patient or a parent with Visual Analogic Scale (froom 0 point = worst to 10 points = best),
  4. sedimentation rate (from 0 to 10).
Evaluation of the physical activity level | Weeks 13, 25 and 49
  The difference of the medium physical activity level is assessed by the continue measures (for 7 days) of the time spent in the MVPA (Moderate to Vigorous Physical Activity) via actimetry (counts/min).
  Actimetric measurements will be performed before the start of the intervention to determine a value for V0, at 13 weeks (for V1), at 25 weeks (for V2), and at 49 weeks (for V3)
Evaluation of the physical activity level | Each day during 50 weeks
  The difference of the medium physical activity level is assessed by the number of steps estimated by the pedometer watch (only for the experimental group).
  Pedometric measurements will be performed throughout the study but collected one week per month to determine a monthly value.
Quantification of the difference in muscle strength | Weeks 14, 26 and 50
  By dynamometry (Newton)
Evolution of quality of life | Weeks 14, 26 and 50
  Difference of the score obtained in the Pediatric Quality of Life (PedsQL) tool. Score out of 100 for children assess and 100 for parents assess. A high score means a reduced quality of life.
Evolution of functional capacities | Weeks 14, 26 and 50
  Assessment by the questionnaire of the ChildHood Assessment Questionnaire (CHAQ-38) tool. Questionaire's score out of 3, it's a medium of 8 items. A high score means reduced functional capacities.
Evolution of pain | Weeks 14, 26 and 50
  Assessment by the Visual Analogic Scale (VAS) of the CHAQ-38 tool. VAS are out of 10. A high score means an increased pain.
Evolution of fatigue | Weeks 14, 26 and 50
  Difference of the score obtained in the PedsQL-Multidimensional Fatigue Scale questionnaire. Score out of 100 for children assess and 100 for parents assess. A high score means a increased fatigue.
Assessment of the feasibility of the program | week 2 to 13
  Assessment of program participation. Participation is the proportion of subjects who agree to participate in the study among eligible patients.
Assessment of the feasibility of the program | week 2 to 13
  Assessment of program completion. Completion is the proportion of subjects who complete the program and proportion of subjects who complete the exercise sessions.
Assessment of the feasibility of the program | week 2 to 13
  Assessment of program adherence. Adherence is the proportion of sessions attended by subjects.
Assessment of the feasibility of the program | week 2 to 13
  Assessment of program compliance. Compliance is the proportion of prescribed exercise during the session actually performed.
Assessment of the feasibility of the program | week 1 to 50
  Assessment of pedometer watch wearing time over the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Claire BALLOT-SCHMIT, MD, Principal Investigator — CHU de Besançon
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - Hospices Civils de Lyon, Lyon
  - Hôpital Nord Franche-Comté, Trévenans

REFERENCES:
- [Derived] Py S, Maylie F, Parmentier AL, Vidal C, Cuinet B, Mauny F, Lohse A, Toussirot E, Yoshimasa S Jr, Tordi N, Binda D, Ballot-Schmit C. ATHLETIQUE: interest of an adapted physical activity program in patients with juvenile idiopathic arthritis: a feasibility and preliminary effectiveness study. Front Immunol. 2023 Jun 27;14:1213799. doi: 10.3389/fimmu.2023.1213799. eCollection 2023. PMID 37441067